CLINICAL TRIAL: NCT03345797
Title: A Multicenter, Open Label, Variable Dose, Two Arm Pilot Paediatric Phase 1 PK Study to Evaluate Testosterone Nasal Gel (4.5% w/w) in Hypogonadal Boys
Brief Title: Evaluation of Testosterone Nasal Gel in Hypogonadal Boys
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of patients and commercial reasons
Sponsor: Acerus Biopharma Inc. (Industry)
Responsible Party: Sponsor
Organization: Acerus Pharmaceuticals Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NAT-2017-01
Record Dates: First submitted 2017-10-10; First posted 2017-11-17 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Hypogonadism
Keywords: Paediatric
MeSH Terms: conditions — Hypogonadism | interventions — Natesto

STUDY DESIGN:
Intervention Model Description: dual arm: naïve vs TRT experienced
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naive patients - ARM 1 (Experimental): TRT naïve subjects, Tanner Stage of 0, receiving Testosterone Nasal Gel [Natesto] - Single dose of 5.5 mg Natesto on Day 1 and a single dose of 11 mg Natesto on Day 2
  Interventions: Drug: Testosterone Nasal Gel [Natesto]
- Non-naive patients - ARM 2 (Experimental): TRT non-naïve subjects (have had prior testosterone treatment), Tanner Stage >/= 3, receiving Testosterone Nasal Gel [Natesto] - Single dose of 11 mg Natesto on Day 1. On Day 2, 11 mg dose of Natesto in the morning and 11 mg dose of Natesto 12 hours later
  Interventions: Drug: Testosterone Nasal Gel [Natesto]

INTERVENTIONS:
Drug: Testosterone Nasal Gel [Natesto] — nasal gel containing 4.5% w/w testosterone

SUMMARY:
PK study to evaluate serum levels of testosterone post nasal delivery in two cohorts of hypogonadal boys.

DETAILED DESCRIPTION:
ARM 1 - 10 prepubertal, 12-17 years old boys with no prior exposure to TRT will receive single dose of 5.5 mg on day one and single dose of 11 mg on day 2 with repeat blood draws to assess serum levels of testosterone and metabolites.

ARM 2 - 10 Tanner Stage 3, 12-17 years old boys on TRT with bone age >= 13 years will receive single dose of 11 mg on day one, and single dose of 11 mg in the morning and a second 11 mg dose in the afternoon on day 2 with repeat blood draws to assess serum levels of testosterone and metabolites.

ELIGIBILITY:
Inclusion Criteria:

ARM 1 (naïve patients): Participants who meet all of the following inclusion criteria will be eligible for participation in the study:

1. Hypogonadal boys;
2. Chronological age 12 to <18 years;
3. No prior exposure to TRT;
4. Prepubertal
5. Parent/guardian and patient able to understand and provide signed informed consent;

ARM 2 (non-naïve patients): Participants who meet all of the following inclusion criteria will be eligible for participation in the study:

1. Hypogonadal boys with a bone age of ≥13 years (a historical value within the last 12 months will be acceptable);
2. Chronological age 12 to <18 years;
3. Taking an existing TRT treatment dose;
4. Tanner Stage ≥3
5. Parent/guardian and patient able to understand and provide signed informed consent;

Exclusion Criteria:

ARM 1 (naïve patients) AND ARM 2 (non-naïve patients): Participants who meet any of the following criteria will be excluded from participation in the study:

1. Any active allergic condition or presentation of symptoms including allergic rhinitis;
2. An upper respiratory tract infection;
3. Use of any form of intranasal medication delivery other than periodic short-term (less than 3 days) use of sympathomimetic decongestants, within the last 3 months;
4. In the opinion of the Investigator, significant intercurrent disease of any type, in particular liver, kidney, heart disease, stroke, or psychiatric illness;
5. History of pituitary or hypothalamic tumors or history of any malignancy excluding basal cell or squamous cell carcinoma of the skin curatively treated by surgery;
6. History of nasal disorders, nasal or sinus surgery, nasal fracture within the previous 6 months or nasal fracture that caused a deviated anterior nasal septum surgery, mucosal inflammatory disorders, specifically Sjogren's syndrome;
7. History of severe adverse drug reactions to testosterone therapies;
8. Current treatment with other androgens (e.g., dehydroepiandrosterone [DHEA]), anabolic steroids, or other sex hormones;
9. Treatment with estrogens, gonadotropin-releasing hormone (GnRH) agonists, or growth hormone within the previous 12 months;
10. Treatment with drugs that interfere with the metabolism of testosterone, such as anastrozole, clomiphene, dutasteride, finasteride, flutamide, ketoconazole, spironolactone, or testolactone;
11. Diabetes mellitus;
12. Participation in any other research study during the conduct of this study or 30 days prior to the initiation of this study.

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — hypogonadal boys
Enrollment: 8 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 48 hours (approx)
  Cmax for serum testosterone, serum DHT and serum estradiol
Area under the curve (AUC) | 48 hours (approx)
  AUC for serum testosterone, serum DHT and serum estradiol
Minimum serum concentration (Cmin) | 48 hours (approx)
  Cmin for serum testosterone, serum DHT and serum estradiol
Time to reach maximum plasma concentration (tmax) | 48 hours (approx)
  tmax for serum testosterone, serum DHT and serum estradiol

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety) | 5 days
  Safety assessments will include adverse events, clinical laboratory measurements of serum testosterone, DHT and estradiol levels, and vital sign measurements. A phone call will be made 3 days after the patient leaves the clinic to collect any SAEs or AEs that may occur.
Incidence of Treatment-Emergent Adverse Events (Tolerability) | 48 hours (approx)
  To include a adverse events that relate to tolerability and a patient and healthcare provider questionnaire on ease of use dispenser and gel administration

CONTACTS AND LOCATIONS:
Overall Officials: Syed Faisal Ahmed, MD, Principal Investigator — Royal Hospital for Children, U. of Glasgow
Locations (3):
- United Kingdom (3):
  - University of Glasgow, Royal Hospital for Children, Glasgow, Scotland
  - Cambridge University Hospital's NHS Foundation Trust, Cambridge
  - Alder Hey Children's Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: No